CLINICAL TRIAL: NCT05566171
Title: The Effect of Probiotic Supported Yogurt Consumption on Gastrointestinal Symptoms Among People Aged 19-64 Years
Brief Title: The Effect of Probiotic Supported Yogurt Consumption on Gastrointestinal Symptoms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: My colleague did not want to continue the study
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Nezire İnce, Asst. Prof., Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0179
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Dysfunction
Keywords: probiotic, gastrointestinal symptoms, constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will be just follow-up for 4 weeks without any intervention
- Interventional Group (Experimental): This group will consume 125 g plain Activia Probiotic Yogurt without any aroma/fruit during 4 weeks/1 month
  Interventions: Dietary Supplement: Activia Probiotic Yogurt

INTERVENTIONS:
Dietary Supplement: Activia Probiotic Yogurt — Activia probiotic Yogurt will be consumed by participants in this group
  Arms: Interventional Group

SUMMARY:
Probiotics have beneficial effect on Gastrointestinal Symptoms. The aim of this study is to determine the effect of probiotic yogurt consumptions on the people who have gastrointestinal symptoms mainly constipation.

DETAILED DESCRIPTION:
In the beginning of the study Constipation Severity Scale and Bristol Stool Scale was applied to the all people who accepted to participate in this study. According to the student T test analysis (α= 0.05, β=0.20 ) 102 people with gastrointestinal symtoms should be included in the study. When 102 people are found with gastrointestinal symptoms second stage of the study will begin. In this stage of the study 102 people are randomly divided into 2 homogeneous groups. 3 day food record will be taken from 102 people at the beginning and again at the end of the study. Probiotic yogurt (Activia Probiotic Yogurt without any aroma-125 g) will be given to one group for 1 month and nothing will be given to the other group (control group).

ELIGIBILITY:
Inclusion Criteria:

* Living in Izmir
* Individuals who are having BMI between 18.5-24.9 kg / m2
* Having gastrointestinal symptoms according to Constipation Severity Scale and Bristol Stool Scale

Exclusion Criteria:

* Having diagnosed gastrointestinal disease
* Regular consumption of probiotic
* Using of drug that affects gastrointestinal system
* Presence of mental illness

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
The severity of gastrointestinal symptoms (mainly constipation) will decrease in the interventional group | 4 weeks
  We expect to see improvement in the gastrointestinal symptoms after consuming probiotic yogurt

CONTACTS AND LOCATIONS:
Overall Officials: Nezire Ince, Study Director — Eastern Mediterranean University
Locations (1):
- Nezire, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No